CLINICAL TRIAL: NCT01121133
Title: A Phase I Study to Assess the Effect of a CYP3A Inducer (Rifampin) on the Pharmacokinetics of ABT-263 (Navitoclax)
Brief Title: A Study to Assess the Effect of Rifampin on the Metabolism of Navitoclax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Kyle Holen, M.D./Medical Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-955
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2011-05

CONDITIONS: Lymphoma, Including Chronic Lymphocytic Leukemia; Solid Tumors
MeSH Terms: conditions — Lymphoma | interventions — navitoclax; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (navitoclax and rifampin) (Experimental)
  Interventions: Drug: navitoclax; Drug: Rifampin

INTERVENTIONS:
Drug: navitoclax — Subjects will be dosed with Navitoclax, then dosed with Navitoclax in combination with Rifampin.
  Other Names: ABT-263, navitoclax
Drug: Rifampin — Subjects will be dosed with Navitoclax, then, dosed with Navitoclax in combination with Rifampin.

SUMMARY:
This is an open-label, single or multiple center study to determine the interaction of rifampin with navitoclax (ABT-263) in approximately 12 subjects with cancer.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older.
* Has a non-hematologic malignancy (radiographic, histologic, or cytologic confirmation), or hematologic malignancy (histologic or cytologic confirmation) that is either: relapsed or refractory to standard therapy, failed at least one prior therapy or no known effective therapy exists.
* In the investigator's opinion, the subject's life expectancy is at least 90 days.
* If clinically indicated, (e.g., subjects over the age of 70) subjects must have documented brain imaging (MRI or CT) negative for subdural or epidural hematoma within 28 days prior to the first dose of study drug.

Exclusion Criteria

* Subjects with brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.
* History of or is clinically suspicious for cancer-related central nervous system (CNS) disease.
* Has undergone an allogeneic stem cell transplant.
* Has an underlying, predisposing condition of bleeding or currently exhibits signs of bleeding.
* Has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Has active immune thrombocytopenic purpura or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
* Significant history of cardiovascular disease (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease. Female subject is pregnant or breast-feeding.
* History of or an active medical condition(s) that affects absorption or motility (e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, etc).
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * tuberculosis
  * diagnosis of fever and neutropenia within 1 week prior to study drug administration
* Received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal (with the exception of hormones for hypothyroidism or estrogen replacement therapy [ERT], or agonists required to suppress serum testosterone levels [e.g., LHRH, GnRH, etc.] for subjects with prostate cancer Subject is currently receiving or requires anticoagulation therapy (e.g., warfarin at any dose) or any drugs or herbal supplements that affect platelet function, with the exception of low-dose heparin used to maintain the patency of a catheter.
* Subject has used known inhibitors (e.g., ketoconazole) or inducers (e.g., rifampin and carbamazepine) of cytochrome P450 3A (CYP3A) within 1 week prior to first dose of study.
* Subject has a history of hypersensitivity to any of the rifamycins.
* In the opinion of the Investigator, the subject is an unsuitable candidate to receive ABT-263.
* History of or is clinically suspicious for cancer-related central nervous system (CNS) disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the effect of rifampin on the pharmacokinetics of navitoclax. | Weekly

SECONDARY OUTCOMES:
To determine the safety of navitoclax when administered alone and in combination with rifampin in these patients. | Daily

REFERENCES:
- [Result] Yang J, Pradhan RS, Rosen LS, Graham AM, Holen KD, Xiong H. Effect of rifampin on the pharmacokinetics, safety and tolerability of navitoclax (ABT-263), a dual inhibitor of Bcl-2 and Bcl-XL , in patients with cancer. J Clin Pharm Ther. 2014 Dec;39(6):680-4. doi: 10.1111/jcpt.12193. Epub 2014 Jul 22. PMID 25047139